CLINICAL TRIAL: NCT06549790
Title: A Phase Ia/Ib Study of NMS-03597812 in Adult Patients With Relapsed/Refractory Acute Myeloid Leukemia Including Patients With TP53 Mutations
Brief Title: Study of NMS-03597812 in Adult Patients With Relapsed/Refractory Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nerviano Medical Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PERKA-812-003
Record Dates: First submitted 2024-07-25; First posted 2024-08-12 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Relapsed/Refractory Acute Myeloid Leukemia
Keywords: Leukemia; Relapsed/Refractory Acute Myeloid Leukemia; TP53 mutations
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NMS-03597812 (Experimental): Dose escalation (Phase Ia):
  Administered orally once daily (28 consecutive days) in repeated 4-week cycles. Each cycle is 28 days.
  Expansion cohorts (Phase Ib, Cohorts A and B):
  The dose expansion may comprise up to a total of 2 single arms of NMS-03597812 as single agent:
  * Cohort A: in patients with TP53mt relapsed/refractory acute myeloid leukemia (R/R AML) prior unfit to intensive chemotherapy (IC) who have exhausted standard treatment options
  * Cohort B: in prior fit or unfit patients to IC with TP53wt R/R AML who have exhausted standard treatment options
  Backfill cohorts:
  Optional backfill cohorts may be opened at any time during the conduct of the trial to further evaluate the following items: NMS-03597812 dosing alone, pharmacokinetic (PK), drug-drug interactions, food effects, biomarkers and QTc for NMS-03597812 as single agent.
  Interventions: Drug: NMS-03597812

INTERVENTIONS:
Drug: NMS-03597812 — Route of Administration: Oral

SUMMARY:
The aim of PERKA-812-003 study is to investigate the safety, pharmacokinetics and preliminary anti-tumor activity of treatment with NMS-03597812 as single agent in Relapsed/Refractory Acute Myeloid Leukemia (R/R AML) patients who have exhausted standard treatment, including a subset of patients with TP53 mutations. It is anticipated that combination with venetoclax will be further evaluated following a future protocol amendment, once the Recommended Range Dose (RDR) as single agent has been defined.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of refractory/relapsed (R/R) AML according to 2022 ELN recommendation:

Phase Ia

* single agent dose escalation of NMS-03597812: R/R AML patients who have exhausted standard therapy: a) prior fit patients to intensive chemotherapy (IC): failed at least one cycle of IC in front-line therapy or b) prior unfit to IC: failed at least 2 cycles of hypomethylating agents (HMA)/venetoclax combination therapy, or at least 4 cycles of HMA monotherapy; c) patients must have failed all other approved therapies for which they are eligible, including FLT3 inhibitors, IDH1/2 inhibitors, and CD33 directed therapy

Phase Ib

* Cohort A: single agent in R/R AML TP53mt patients who have exhausted standard therapy: a) prior unfit to intensive chemotherapy (IC): failed at least 2 cycles of HMA/venetoclax combination therapy, or at least 4 cycles of HMA monotherapy; b) patients must have failed all other approved therapies for which they are eligible, including FLT3 inhibitors, IDH1/2 inhibitors, and CD33 directed therapy
* Cohort B: single agent in R/R AML TP53wt patients who have exhausted standard therapy: a) prior fit patients to intensive chemotherapy (IC): failed at least one cycle of IC in front-line therapy or b) prior unfit to IC: failed at least 2 cycles of HMA/venetoclax combination therapy, or at least 4 cycles of HMA monotherapy; c) patients must have failed all other approved therapies for which they are eligible, including FLT3 inhibitors, IDH1/2 inhibitors, and CD33 directed therapy
* Adult (age ≥ 18 years) patients
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Unless agreed with sponsor, the interval from prior antitumor treatment should be at least 2 weeks or 5 half-lives, whichever is longer, other than hydroxyurea
* All acute toxic effects (excluding alopecia) of any prior therapy must have resolved to NCI CTCAE version 5.0 Grade≤ 1
* Adequate organ function
* Must use highly effective contraception or true abstinence. Female patients must be surgically sterile or, if patient is of childbearing potential, must agree to use effective contraception of therapy and in the following 210 days after discontinuation of study treatment. Since NMS-03597812 has potential induction of CYP3A4, women of childbearing potential must be advised that hormonal contraceptives might lose efficacy and must use alternate form of highly effective contraception. Male patients must be surgically sterile or must agree to use highly effective contraception or true abstinence during the period of therapy and in the following 120 days for male patients who must refrain from donating sperm during this period after discontinuation of study treatment.
* Capability to swallow capsules intact (without chewing, crushing, or opening)
* Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests and other study indications or procedures
* Signed and dated Independent Ethics Committee (IEC) or Institutional Review Board (IRB)-approved informed consent form indicating that the patient is aware of the neoplastic nature of his/her disease and has been informed of the procedures to be followed, the investigational nature of the therapy, potential benefits, side effects, discomforts, risks, and alternative treatments.

Exclusion Criteria:

* Current enrollment in another interventional clinical study unless only participating in survival follow up
* White blood cells (WBC) count >20×10^3/microliter (μL). However, patients can be treated with hydroxyurea and/or leukapheresis prior to study treatment start to reduce the WBC to ≤ 20×10^3/μL to enable eligibility for study drug dosing.
* Diagnosis of acute promyelocytic leukemia or BCR-ABL-positive leukemia
* Currently active second malignancy, except for adequately treated basal or squamous cell skin cancer and/or cone biopsied in situ carcinoma of the cervix uteri and/or superficial bladder cancer.
* Patients with known leukemia involvement of central nervous system (CNS).
* Hematopoietic stem cell transplantation (HSCT) within 3 months of treatment start and/or persistent non- hematologic toxicities of Grade ≥2 related to the transplant
* Active acute or chronic graft versus host disease (GVHD) requiring immunosuppressive treatment
* Patients with QTcF interval ≥ 470 milliseconds or with risk factors for torsade de pointes (e.g., uncontrolled heart failure, uncontrolled hypokalemia, history of prolonged QTc interval or family history of long QT syndrome). For patients receiving treatment with concomitant medications known to prolong the QTc interval, replacement with another treatment needs to be considered. If replacement or discontinuation is not clinically feasible, a careful risk/benefit evaluation should be performed prior to enrollment.
* Pregnancy. All female patients with reproductive potential must have a negative pregnancy test (serum or urine) within the screening period prior to start of study drug.
* Breast-feeding or planning to breast feed during the study or within 90 days after study treatment.
* Known active gastrointestinal disease (eg, gastro-duodenal ulcer, gastrectomy, Crohn's disease, ulcerative colitis, or short gut syndrome) or other malabsorption syndromes that would impact on drug absorption.
* Patient who are receiving concomitant medications with antacids (proton pump inhibitors are strictly prohibited; calcium carbonate antacids are only allowed 6 hours prior to a dose or 1 hour after). Note: exclusion criterion not applicable to optional backfill cohort for investigation of drug-drug interaction with antiacids.
* Patient who are receiving concomitant medications that are strong inducers or inhibitors of CYP3A4 (with the exception of azole antifungals) and CYP2C9 that cannot be replaced with alternative therapy.
* Patients who are receiving concomitant medications that are sensitive substrates of CYP3A4,CYP2D6, CYP1A2 and CYP2B6 with narrow therapeutic window that cannot be replaced with alternative therapy. Drugs with broad therapeutic indices may still be acceptable.
* Patients who are receiving concomitant medications that are strong or moderate P-gp inhibitors that cannot be replaced with alternative therapy.
* Major surgery within 4 weeks before study treatment start.
* Radiotherapy within 4 weeks before study treatment start. However, if the radiation portal covered ≤5 % of the bone marrow reserve, the patient may be enrolled irrespective of the end date of radiotherapy.
* History of necrotic pancreatitis or acute severe pancreatitis, requiring medical intervention and/or hospitalization, in the previous 6 months before study treatment start.

NOTE: Other protocol defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2024-10-16 (Actual); Primary Completion 2029-09-15 (Estimated); Study Completion 2030-05-15 (Estimated)

PRIMARY OUTCOMES:
Phase Ia (escalation) - Number of Participants with Adverse Events (AEs) | Screening (Day ≤28) up to 28-day follow-up after end of treatment (Approximately 13 months)
  Evaluation of AE frequency and severity (graded using the National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] Version 5.0), including dose limiting toxicities (DLTs), laboratory measurements, electrocardiogram (ECG) measurements, vital sign measurements
Phase Ib (expansion) - Complete Remission (CR) rate | From date of treatment initiation up to hematological relapse (Approximately 12 months)
  Complete Remission (CR) rate, as defined by the Investigators based on the 2022 European LeukemiaNet (ELN) recommendations

SECONDARY OUTCOMES:
Phase Ia - Complete remission (CR) rate | From date of treatment initiation up to hematological relapse (Approximately 12 months)
  Complete Remission (CR) rate, as defined by the Investigators based on the 2022 European LeukemiaNet (ELN) recommendations.
Phase Ia - Maximum concentration (Cmax) of NMS-0597812 | Cycle 1 (each cycle is 28 days): Day 1 and Day 15
  Plasma samples will be collected and used for pharmacokinetics assessments
Phase Ia - Related time of achievement of occurrence of Cmax (tmax) of NMS-0597812 | Cycle 1 (each cycle is 28 days): Day 1 and Day 15
  Plasma samples will be collected and used for pharmacokinetics assessments
Trough concentration (Cτ) area under concentration versus time up to 24 hours (dosing interval) of NMS-0597812 | Cycle 1 (each cycle is 28 days): Day 1 and Day 15
  Plasma samples will be collected and used for pharmacokinetics assessments
Phase Ia - Half-life of the terminal phase (t½,z) of NMS-0597812 | Cycle 1 (each cycle is 28 days): Day 1 and Day 15
  Plasma samples will be collected and used for pharmacokinetics assessments
Phase Ia - Plasma clearance (CL) of NMS-0597812 | Cycle 1 (each cycle is 28 days): Day 1 and Day 15
  Plasma samples will be collected and used for pharmacokinetics assessments
Phase Ia - Volume of distribution (Vss) of NMS-0597812 | Cycle 1 (each cycle is 28 days): Day 1 and Day 15
  Plasma samples will be collected and used for pharmacokinetics assessments
Phase Ia - Accumulation ratio (Rac) of NMS-0597812 | Cycle 1 (each cycle is 28 days): Day 15
  Plasma samples will be collected and used for pharmacokinetics assessments
Phase Ia - Renal clearance (CLR) of NMS-03597812 excreted in urine (data permitting) | Cycle 1 (each cycle is 28 days): Day 1 and Day 15
  Urine samples will be collected and used for pharmacokinetics assessments
Phase Ia - Cumulative amount recovered unchanged in the urine (Ae) of NMS-03597812 (data permitting) | Cycle 1 (each cycle is 28 days): Day 1 and Day 15
  Urine samples will be collected and used for pharmacokinetics assessments
Phase Ia - Cumulative amount recovered unchanged in the urine expressed as a fraction of administered dose (Ae%) of NMS-03597812 (data permitting) | Cycle 1 (each cycle is 28 days): Day 1 and Day 15
  Urine samples will be collected and used for pharmacokinetics assessments
Phase Ib - Complete remission (CR) + complete remission with partial hematologic recovery (CRh) rate | From date of treatment initiation up to hematological relapse (Approximately 12 months)
  Number and percentage of patients who achieve CR and CRh as best response
Phase Ib - Complete remission (CR) + Complete remission with incomplete hematologic recovery (CRi) rate | From date of treatment initiation up to hematological relapse (Approximately 12 months)
  Number and percentage of patients who achieve CR and CRi as best response
Phase Ib - Complete remission (CR) + Complete remission with partial hematologic recovery (CRh) + complete remission with incomplete hematologic recovery (CRi) rate | From date of treatment initiation up to hematological relapse (Approximately 12 months)
  Number and percentage of patients who achieve CR, CRh and CRi as best response
Phase Ib - Overall Response Rate (ORR: CR + CRh + CRi + MLFS + PR) | From date of treatment initiation up to hematological relapse/progressive disease (Approximately 12 months)
  ORR: Complete remission (CR) + Complete remission with partial hematologic recovery (CRh) + Complete remission with incomplete hematologic recovery (CRi) + Morphological leukemia-free state (MLFS) + Partial remission (PR)
  Defined as the number and percentage of patients who achieve CR, CRh, CRi, MLFS and PR as best response in the analysis population
Phase Ib - Overall Survival (OS) | First dose to the date of death from any cause or start of a new anti-cancer therapy, whichever comes first (Approximately 18 months)
  Defined as the time from the date of start of treatment until the date of death from any cause. Patient who was not known to have died by the end of study will be censored at the date of last recorded date.
Phase Ib - Duration of Response (DoR) | From the date of first response (CR, CRh, or CRi) to the date of hematological relapse or death due to progression, whichever comes first. (Approximately 12 months)
  Defined as the time from the date of first response (CR, CRh, or CRi) until the date of documented hematologic relapse or death due to progression. DOR will be also calculated for overall response, including patients who achieve MLFS or PR as best response during the treatment.
Phase Ib - Event-Free Survival (EFS) | From the date of treatment initiation to the date of hematological relapse from CR, CRh, or CRi, date of treatment failure, or death from any cause, whichever comes first. (Approximately 18 months)
  Defined as the time from the date of treatment initiation to the date of hematological relapse from CR, CRh, or CRi, or death from any cause, whichever comes first.
Phase Ib - Relapse-free Survival (RFS) | Date of first achievement of remission until the date of hematologic relapse or death from any cause, whichever comes first (Approximately 12 months).
  Measured only for patients achieving CR, CRh, or CRi, and it is defined as the time from the date of first achievement of remission until the date of hematologic relapse or death from any cause.
Phase Ib - Proportion of patients bridged to hemopoietic stem cell transplantation (HSCT) | From date of treatment initiation up to end of study (Approximately 18 months)
Phase Ib - Rate of conversion from transfusion-dependence to transfusion independence | From date of treatment initiation up to end of study (Approximately 18 months)
Phase Ib - AE frequency and severity | Screening (Day ≤28) up to 28-day follow-up after end of treatment (Approximately 13 months)
  AE frequency and severity (graded using the National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] Version 5.0), laboratory, ECG and vital sign measurements

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - City of Hope - Duarte, Duarte, California
  - Rocky Mountain Cancer Centers, Aurora, Colorado
  - Medical Oncology Hematology Consultants, Newark, Delaware
  - Blood and Marrow Transplant Group of Georgia, Atlanta, Georgia
  - Mayo Clinic Cancer Center (MCCC) - Rochester, Rochester, Minnesota
  - Gabrail Cancer Research Center, Canton, Ohio
  - The University of Texas MD Anderson Cancer Center, Houston, Texas